CLINICAL TRIAL: NCT01420510
Title: Saginil in Vaginal Cannulas vs. Placebo for the Prevention of Vaginitis in Gynecologic Oncologic Patients Receiving Chemotherapy: a Randomized Controlled Trial.
Brief Title: Saginil in vs. Placebo for Gynecologic Oncology Patients Affected by Vaginitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Fabio Ghezzi, Professor, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Saginil in vaginitis
Record Dates: First submitted 2011-08-16; First posted 2011-08-19 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Vaginitis
Keywords: Patients satisfaction; Side effects
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adelmidrol (Experimental): Efficacy of Adelmidrol vaginal gel in preventing vaginitis in oncologic patients
  Interventions: Drug: Adelmidrol vaginal gel
- Placebo (Placebo Comparator): Efficacy of Placebo in preventing vaginitis in oncologic patients
  Interventions: Drug: Placebo vaginal gel

INTERVENTIONS:
Drug: Adelmidrol vaginal gel — Application of a Adelmidrol vaginal gel
  Arms: Adelmidrol
Drug: Placebo vaginal gel — Application of a placebo vaginal gel
  Arms: Placebo

SUMMARY:
We hypothesise that the use of Adelmidrol (Saginil in vaginal cannulas) can reduce the incidence and magnitude of vaginitis in patients affected by gynecologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Gynecologic malignancy
* Current administration of chemotherapy

Exclusion Criteria:

* Colpectomy
* Vaginal cancer
* Vulvar cancer
* Bacterial vaginitis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with vaginitis in the group taking Adelmidrol (vaginal cannulas) vs. number of patients with vaginitis in the Placebo group | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gynecologic Oncology Unit, Varese, Italy